CLINICAL TRIAL: NCT03442972
Title: Investigating the Release of Stored Enteral Lipids in Response to a Single Subcutaneous Dose of Analogue Glucagon-like Peptide-2 in Humans
Brief Title: Glucagon-like Peptide-2 Mediated Secretion of Stored Enteral Lipids
Acronym: GLP-2 Biopsy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Kensington Screening Clinic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-6368.2
Record Dates: First submitted 2018-02-02; First posted 2018-02-22 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2020-11

CONDITIONS: Hyperlipidemias
Keywords: Intestinal lipoprotein; Duodenal biopsy; Gut Peptide; Chylomicrons
MeSH Terms: conditions — Hyperlipidemias | interventions — teduglutide

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to receive either teduglutide or placebo as a single subcutaneous injection, 1 hour prior to duodenal biopsy
Who Masked: Participant
Masking Description: Single-blinded study with participant blinded to treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teduglutide (Experimental): Teduglutide, up to 0.05mg/kg, subcutaneous, single dose
  Interventions: Drug: Teduglutide
- Placebo (Placebo Comparator): Placebo, subcutaneous, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Teduglutide — Teduglutide
  Arms: Teduglutide
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Some of the fat (triglyceride) from the food humans eat gets stored in the bowel. This triglyceride can then be released into the blood when another meal is consumed or in response to hormones. How the gut hormone glucagon-like peptide-2 (GLP-2) releases the triglyceride from the gut is not known. The research team in this study is interested in finding out how teduglutide (a degradation resistant form of GLP-2) releases stored triglyceride from the gut by studying samples from patients undergoing endoscopy and small bowel biopsy.

DETAILED DESCRIPTION:
The release of stored enteral lipids will be investigated in 30 patients undergoing upper gastrointestinal endoscopy and duodenal biopsy for clinical indications. Patients undergoing the procedure will be recruited. Participants will have a high fat liquid meal as breakfast. 5 hours later, participants will be randomly assigned to receive either a subcutaneous injection of placebo (n=15) or a subcutaneous injection of the Health Canada approved glucagon-like peptide-2 (GLP-2) analogue (teduglutide, Revestive®, Shire Canada)(n=15 different subjects). 1 hour later, a duodenal biopsy specimen will be obtained from 2-3 sample sites,snap frozen in dry ice and stored at -80°C for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, aged 18 to 60 years requiring endoscopy and duodenal biopsies for clinical indications, with no contraindications to the procedure, as judged by Dr. Bookman of the Kensington Screening Clinic, Toronto, ON, Canada

Exclusion Criteria:

* Patients with active inflammatory bowel disease
* Patients with pre-existing Celiac disease, exocrine pancreatic insufficiency or small bowel malabsorption
* Patients with active bowel malignancy
* Patients with diabetes mellitus or known/ suspected motility disorders of the gut
* Patients with decompensated liver disease
* Patients on ezetimibe or bile acid sequestrants
* Patients who are pregnant or breastfeeding.
* Patients with renal disease
* Patients on benzodiazepine
* Unstable cardiac or respiratory disease
* Any changes to medication in the preceding month

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Release of enteral lipids in response to teduglutide | 6 hours
  To quantify the difference in amount of enteral lipids between GLP-2 and placebo treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Lewis, MD, Principal Investigator — UHN
Locations (2):
- Canada (2):
  - Toronto General Hopital, Toronto, Ontario
  - Kensington Screening Clinic, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No